CLINICAL TRIAL: NCT05754060
Title: Cognitive Processing Slowness as a Marker of Cognitive Impairment in Non-central Nervous System Cancer Patients
Acronym: RIVAGE
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220816
Record Dates: First submitted 2023-02-22; First posted 2023-03-03 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer; Colon Cancer; Cognitive Impairment
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Saint-Louis Lille Battery (SSLIB): Saint-Louis Lille Battery (SSLIB) is composed of three tests studying the speed of cognitive processing and proposed to the subjects on a tactile tablet. These three tasks are:
  (a) Reaction time tasks specifically developed for this study b) A digital adaptation of the WAIS-IV code subtest c) A digital version of the Trail Making Test (A and B)
  Interventions: Other: Saint-Louis Lille Battery (SSLIB)

INTERVENTIONS:
Other: Saint-Louis Lille Battery (SSLIB) — Saint-Louis Lille Battery (SSLIB) composed of three tests studying the speed of cognitive processing and proposed to the subjects on a tactile tablet. These three tasks are:
  (a) Reaction time tasks specifically developed for this study b) A digital adaptation of the WAIS-IV code subtest c) A digital version of the Trail Making Test (A and B)

SUMMARY:
Cancer is a frequent disease considering that one person out of three will be confronted with it in their lifetime. Cancer patients often express complaints related to cognitive impairment as an outcome of their oncological treatment. These cognitive disorders have a significant impact on the patient's and their carer's quality of life. Therefore, it appears necessary to have a reliable, quick and simple tool in order to detect cognitive impairment.

The rationale of this study relies on 3 main points :

* The cognitive complaint frequently reported by cancer patients
* The difficulty in reliably demonstrating the cause of this complaint through conventional neuropsychological tests
* The interest of cognitive processing speed as an indicator of cognitive dysfunction

The primary objective of the study is to evaluate a potential variation of cognitive processing speed at the Saint-Louis Lille Battery (SSLIB) between the beginning and during (4 months after the beginning) the oncological treatment of adults with breast cancer or colon cancer.

ELIGIBILITY:
Inclusion Criteria:

* Beginning an oncological treatment for breast or colon cancer
* Patients of age ≥ 20 and ≤ 70 years old
* Cancer diagnosis announcement delivered since less than 3 weeks (+/- a week)
* Patient affiliated to French social security

Exclusion Criteria:

* Patient's opposition to the study
* Notion of an abnormal cerebral scan or MRI
* Drug use (alcohol, narcotics…)
* Chronic (≥ 15 days) treatment with corticosteroids > 1mg/kg/j (prednisone or equivalent)
* Ocular pathology or cognitive disorder impairing comprehension and reading abilities
* Patients under curatorship, guardianship or under the protection of justice

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients with breast cancer or colon cancer
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients for which there is a variation of reaction time between the beginning and during the oncological treatment at M4 | At 4 months
  The variation will be defined as follows :
  * Mild if the reaction times vary for only one of the Saint-Louis Lille Battery (SLLIB) tests
  * Moderate if the variation appears on two of the SLLIB tests
  * Severe if the variation appears on three of the SLLIB tests

SECONDARY OUTCOMES:
Proportion of patients for which there is a variation of reaction time between the beginning and after the end of the oncological treatment (M12) | At 12 months
  The variation will be defined as follows :
  * Mild if the reaction times vary for only one of the Saint-Louis Lille Battery (SLLIB) tests
  * Moderate if the variation appears on two of the SLLIB tests
  * Severe if the variation appears on three of the SLLIB tests
Proportion of patients for which there is a variation of reaction time between M4 and M12 | At 12 months
  The variation will be defined as follows :
  * Mild if the reaction times vary for only one of the Saint-Louis Lille Battery (SLLIB) tests
  * Moderate if the variation appears on two of the SLLIB tests
  * Severe if the variation appears on three of the SLLIB tests
Anxiety and depression levels | At inclusion
  Anxiety and depression levels will be assessed using the Hamilton Anxiety Depression scale : The HAD scale is a self-assessment scale for detecting states of depression and anxiety in the setting of an hospital medical outpatient clinic.
  HADS is a self-administered scale of 14 items which assessed levels of depression and anxiety, divided into 2 subscales of 7 items (Anxiety or HADS-A, Depression or HADS-D). Each item is scored on a scale of 0 to 3. A score is generated for each of the two sub-scales (sum of the 7 items, ranging from 0 to 21). Limit scores, for each of the scores, distinguish: non-cases or asymptomatic ones (score ≤ 7); probable or borderline cases (score 8-10); clearly or clinically symptomatic cases (score ≥ 11).
Anxiety and depression levels | At 4 months
  Anxiety and depression levels will be assessed using the Hamilton Anxiety Depression scale : The HAD scale is a self-assessment scale for detecting states of depression and anxiety in the setting of an hospital medical outpatient clinic.
  HADS is a self-administered scale of 14 items which assessed levels of depression and anxiety, divided into 2 subscales of 7 items (Anxiety or HADS-A, Depression or HADS-D). Each item is scored on a scale of 0 to 3. A score is generated for each of the two sub-scales (sum of the 7 items, ranging from 0 to 21). Limit scores, for each of the scores, distinguish: non-cases or asymptomatic ones (score ≤ 7); probable or borderline cases (score 8-10); clearly or clinically symptomatic cases (score ≥ 11).
Anxiety and depression levels | At 12 months
  Anxiety and depression levels will be assessed using the Hamilton Anxiety Depression scale : The HAD scale is a self-assessment scale for detecting states of depression and anxiety in the setting of an hospital medical outpatient clinic.
  HADS is a self-administered scale of 14 items which assessed levels of depression and anxiety, divided into 2 subscales of 7 items (Anxiety or HADS-A, Depression or HADS-D). Each item is scored on a scale of 0 to 3. A score is generated for each of the two sub-scales (sum of the 7 items, ranging from 0 to 21). Limit scores, for each of the scores, distinguish: non-cases or asymptomatic ones (score ≤ 7); probable or borderline cases (score 8-10); clearly or clinically symptomatic cases (score ≥ 11).
Cognitive complaint | At inclusion
  Cognitive complaint will be assessed using the Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) questionnaire v3.
  It is made up 37 items divided in four subscales: perceived cognitive impairments (PCI); perceived cognitive abilities ; impact of perceived cognitive impairment on Quality Of Life; and comments from others on cognitive function. It ranges from 0 to 148. The higher the score, the better the cognitive function.
Cognitive complaint | At 4 months
  Cognitive complaint will be assessed using the Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) questionnaire v3.
  It is made up 37 items divided in four subscales: perceived cognitive impairments (PCI); perceived cognitive abilities ; impact of perceived cognitive impairment on Quality Of Life; and comments from others on cognitive function. It ranges from 0 to 148. The higher the score, the better the cognitive function.
Cognitive complaint | At 12 months
  Cognitive complaint will be assessed using the Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) questionnaire v3.
  It is made up 37 items divided in four subscales: perceived cognitive impairments (PCI); perceived cognitive abilities ; impact of perceived cognitive impairment on Quality Of Life; and comments from others on cognitive function. It ranges from 0 to 148. The higher the score, the better the cognitive function.
Quality of life assessed with the QLQ-C30 questionnaire | At inclusion
  Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30- v3). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
Quality of life assessed with the QLQ-C30 questionnaire | At 4 months
  Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30- v3). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
Quality of life assessed with the QLQ-C30 questionnaire | At 12 months
  Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30- v3). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.

IPD SHARING:
Plan to Share IPD: Undecided